CLINICAL TRIAL: NCT02100280
Title: A Double-blinded, Randomized, Parallel Design Study to Compare the Effect of Deep Block Versus Moderate Block on the Stress Response After Laparoscopic Gastrectomy
Brief Title: The Effect of Deep Block Versus Moderate Block on the Stress Response After Laparoscopic Gastrectomy
Acronym: suga-SH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, BON WOOK KOO, assistant professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SNUBH-NMB
Record Dates: First submitted 2014-03-23; First posted 2014-03-31 (Estimated); Results first posted 2018-05-21 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Neuromuscular Blockade
Keywords: Neuromuscular blockade; Sugammadex; Laparoscopic surgery; IL-6
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- deep block (Experimental): After induction of anesthesia, continuous neuromuscular monitoring is started after calibration and stabilization of the signal as recommended by good clinical research practice; 50 Hz tetanic stimulation for 5 s, calibration, stabilization for at least 2 min 2. After stabilization, rocuronium 0.6 mg/kg is administered IV within 5 s for tracheal intubation. Maintenance dose of 0.1-0.2 mg/kg rocuronium is administered as needed for the maintenance of post tetanic count 1-2 (deep block). At the end of surgery, sugammadex 4 mg/kg are administered IV for reversal of neuromuscular block.
  Interventions: Drug: deep block
- moderate block (No Intervention): After induction of anesthesia, continuous neuromuscular monitoring is started after calibration and stabilization of the signal as recommended by good clinical research practice; 50 Hz tetanic stimulation for 5 s, calibration, stabilization for at least 2 min 2. After stabilization, rocuronium 0.6 mg/kg is administered IV within 5 s for tracheal intubation. Maintenance dose of 0.1-0.2 mg/kg rocuronium is administered as needed for the maintenance of train of four count 1-2 (moderate block). At the end of surgery neostigmine 50 ㎍/kg with glycopyrrolate 10 ㎍/kg are administered IV for reversal of neuromuscular block.

INTERVENTIONS:
Drug: deep block — sugammadex 4 mg/kg are administered IV for reversal of neuromuscular block
  Other Names: bridion
  Arms: deep block

SUMMARY:
This study is a multicenter, randomized, controlled, double-blinded, and parallel design study. A total of 96 patients were decided to be recruited considering a 10% dropout rate. Patients are randomized to receive a deep block or a moderate block. The randomization numbers are generated using a computer-generated randomization code (1) and are sealed in the opaque envelope until they are handed over to the anesthesiologist in charge of anesthesia management after the induction of anesthesia. Patients, surgeons reporting the scale of surgical status, and another researcher analysing the cytokines levels are blinded to the patient group. Patients aged 18-65 yr, ASA 1 or 2, and are scheduled for elective laparoscopic gastrectomy are included. Patients with severe respiratory or cardiac disease, hepatic or renal function impairment, on medications affecting neuromuscular function, and with known allergy to the drugs to be used are excluded.

DETAILED DESCRIPTION:
Induction and maintenance of anesthesia

Premedication is done with midazolam 0.03 mg/kg IV at reception area. Anesthesia is induced and maintained with intravenous propofol, remifentanil, and rocuronium. The dose of propofol is adjusted to maintain BIS value to 40-60, remifentanil to maintain blood pressure within 20% of preoperative value, and rocuronium to maintain PTC 1-2 (deep block) or TOF1-2 (moderate block). The monitoring consists of ECG, NIBP, pulse oximetry, temperature, ETCO2, BIS, and neuromuscular monitoring with acceleromyography (TOF-Watch SXTM, Organon Ltd., Dublin, Ireland).

Management and monitoring of neuromuscular block

After induction of anesthesia, continuous neuromuscular monitoring is started after calibration and stabilization of the signal as recommended by good clinical research practice; 50 Hz tetanic stimulation for 5 s, calibration, stabilization for at least 2 min 2. After stabilization, rocuronium 0.6 mg/kg is administered IV within 5 s for tracheal intubation. Maintenance dose of 0.1-0.2 mg/kg rocuronium is administered as needed for the maintenance of PTC1-2 (deep block) or TOF1-2 (moderate block). At the end of surgery, sugammadex 4 mg/kg for deep block group or neostigmine 50 ㎍/kg with glycopyrrolate 10 ㎍/kg for moderate block group are administered IV for reversal of neuromuscular block.

Evaluation of surgical conditions

A 5-point surgical rating scale (1 = excellent, 2 = good, 3 = acceptable, 4 = poor, 5 = extremely poor) is rated by the surgeon who is in charge of the patient's operation and is blind to the patient's group assignment. Intraoperative patient movement reported by surgeon, checked by restoration of spontaneous respiration or sudden increase in PIP, and any other movement are also recorded.

Measurement of cytokines and acute phase reactants

Blood samples are collected from the antecubital vein of the arm not used for IV infusion preoperatively, at the end of peritoneal closure, and 1, 2, & 48 hr after the end of operation for analysis of TNF-α, IL-1β, 6, 8 and CRP. The blood samples are collected at test tubes and sent to the laboratory on ice. Cytokines are analyzed with enzyme-linked immunosorbent assay and CRP is determined by an institutional chemistry analyzer.

Postoperative pain measurement

Postoperative pain is evaluated by verbal numerical rating scale (VNRS, 0 = no pain, 10 = the severest pain imaginable) at postoperative 1, 2, 6, 24, and 48 hr. Postoperative pain is controlled by IV patient controlled analgesia using fentanyl. If patient complain of severe pain (VNRS score of 7 or more), additional analgesics can be used according to the attending physician. The amount of fentanyl used and additional analgesic drugs used are reported.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists grade 1 or 2
* Scheduled for elective laparoscopic gastrectomy

Exclusion Criteria:

* Severe respiratory or cardiac disease
* Severe hepatic or renal function impairment
* On medications affecting neuromuscular function
* Known allergy to the drugs to be used

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2014-06-29 (Actual); Primary Completion 2017-06-14 (Actual); Study Completion 2017-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ah-Young Oh, MD.,Ph.D., Study Chair — Seoul national univ. BUNDANG hospital

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Deep Block: Maintenance dose of 0.1-0.2 mg/kg rocuronium is administered as needed for the maintenance of post tetanic count 1-2 (deep block). At the end of surgery, sugammadex 4 mg/kg are administered IV for reversal of neuromuscular block.
- Moderate Block: Maintenance dose of 0.1-0.2 mg/kg rocuronium is administered as needed for the maintenance of train of four count 1-2 (moderate block). At the end of surgery neostigmine 50 ㎍/kg with glycopyrrolate 10 ㎍/kg are administered IV for reversal of neuromuscular block.
Period: Overall Study
Arm/Group | Deep Block | Moderate Block
Started | 48 | 48
Completed | 44 | 44
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deep Block | Moderate Block | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 39 | 73
  >=65 years | 14 | 9 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 34 | 34 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 48 | 48 | 96
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
stress response [Count of Participants; unit: Participants] — Stress response were analyzed Cytokines(TNF-α, IL-1β, IL-6, IL-8, and C-reactive protein) Blood samples were collected from the antecubital vein of the arm not used for IV infusion at preoperatively, at the end of peritoneal closure, and at 2 and 48hrs after the end of operation for analysis of TNF-α, IL-1β, IL-6, IL-8, and C-reactive protein (CRP). Cytokines were analysed with enzyme-linked immunosorbent assay kit(R&D Systems, Minneapolis, Minnesota, USA) and CRP was determined by an institutional chemistry analyser(Beckman Coulter, Brea, Califonia, USA).
  Participants | 44 | 44 | 88

OUTCOME MEASURES:

1. Primary Outcome: IL-6
Description: Blood samples are collected from the antecubital vein of the arm not used for IV infusion 1 hr after the end of operation for analysis of IL- 6.
Time Frame: 1 hr after the end of operation
Measure: Mean (Standard Deviation); unit: pg / ml
Arm/Group | Deep Block | Moderate Block
Number analyzed (Participants) | 44 | 44
pg / ml | 84 (96.98) | 70.14 (99.15)

2. Secondary Outcome: TNF-α
Description: Blood samples are collected from the antecubital vein of the arm not used for IV infusion at the end of peritoneal closure for analysis of TNF-α.
Time Frame: 30min before end of operation
Measure: Mean (Standard Deviation); unit: pg / ml
Arm/Group | Deep Block | Moderate Block
Number analyzed (Participants) | 44 | 44
pg / ml | 1.33 (0.71) | 1.66 (1.75)

3. Secondary Outcome: IL-1β
Description: Blood samples are collected from the antecubital vein of the arm not used for IV infusion at the end of peritoneal closure for analysis of IL-1β.
Time Frame: 30min before end of operation
Measure: Mean (Standard Deviation); unit: pg / ml
Arm/Group | Deep Block | Moderate Block
Number analyzed (Participants) | 44 | 44
pg / ml | 0.34 (0.55) | 0.27 (0.33)

4. Secondary Outcome: IL-8
Description: Blood samples are collected from the antecubital vein of the arm not used for IV infusion 1 hr after the end of operation for analysis of IL- 8.
Time Frame: 1 hr after end of operation
Measure: Mean (Standard Deviation); unit: pg / ml
Arm/Group | Deep Block | Moderate Block
Number analyzed (Participants) | 44 | 44
pg / ml | 29.6 (13.9) | 29.5 (19.4)

5. Secondary Outcome: CRP
Description: Blood samples are collected from the antecubital vein of the arm not used for IV infusion 48 hr after the end of operation for analysis of CRP.
Time Frame: 48 hr after end of operation
Measure: Mean (Standard Deviation); unit: pg / ml
Arm/Group | Deep Block | Moderate Block
Number analyzed (Participants) | 44 | 44
pg / ml | 12.2 (6.4) | 10.6 (5.6)

ADVERSE EVENTS:
Time Frame: adverse event data were not collected
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Deep Block | Moderate Block
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/80/NCT02100280/Prot_SAP_000.pdf